CLINICAL TRIAL: NCT05084287
Title: Robot-assisted and Connected 6-minute Walk Test (TM6)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: PEPPER
Record Dates: First submitted 2021-10-04; First posted 2021-10-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the reliability of the PEPPER robot in assisting and recording the parameters of a TM6. Patients referred to the EFRED service for the performance of a 6MWT will be assisted during their test by the PEPPER robot. The PEPPER robot will also collect the parameters of the 6MWT and produce a report. The EFRED service technician will remain present during the 6MWT and will take note of the test parameters. An evaluation of patient satisfaction with the assistance of the Robot Pepper in the realization of the 6MWT will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Speak fluent French.

Exclusion Criteria:

* Patient's refusal to participate in the study
* Language barrier
* Cognitive disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients referred for 6MWT to the EFRED department of the Pitié Salpêtrière hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
6MWT parameters Robot vs Technician | 1 day
  Measurement of the distance traveled by the patient compared to the measurement made by the medical technician

CONTACTS AND LOCATIONS:
Locations (1):
- AP HP, Paris, France